CLINICAL TRIAL: NCT04477213
Title: Risk Profiling of the Occupational Exposure of COVID-19 to Healthcare Workers- A Multicentric Retrospective Study
Brief Title: Risk Profiling of the Occupational Exposure of COVID-19 to Healthcare Workers.
Status: Completed | Type: Observational
Sponsor: NMC Specialty Hospital (Other)
Responsible Party: Principal Investigator, Prashant Nasa, Specialist Critical Care Medicine, NMC Specialty Hospital
Other Study IDs: NMCHCW-COVID
Record Dates: First submitted 2020-07-17; First posted 2020-07-20 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: COVID19; Healthcare Workers
Keywords: COVID-19; Healthcare Workers; occupational risk of COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose to conduct a retrospective study to define and quantify the variable occupational and non-occupational risk among various HCWs who got COVID-19 . The investigators aim to determine the rates of acquisition of COVID-19, in the context of level of exposure , adequacy of PPE use and other infection control measuresrecommended for COVID-19 and also to define the risk of secondary disease transmission to other household members of HCWs.

DETAILED DESCRIPTION:
Risk of transmission of COVID-19 virus to healthcare workers (HCWs) is matter of debate since the start of this pandemic. In absence of adequate research, the transmission risk is based on non-human studies, non-HCWs epidemiological studies and experiences from previous pandemics or epidemics. The true magnitude of the risk to HCWs has not been clearly estimated. In absence of good scientific data, general recommendations create confusion and mistrust among HCWs. Besides lots of myth and misconceptions among the HCWs including physician adds to emotional and physical challenge in reduction of nosocomial transmission of COVID-19.

COVID-19 related lockdowns have disrupted the global supply-chain and good quality personal protective equipment (PPE) has become an intense matter of discussion from the start of pandemic. The rational use of PPE has become necessity to ensure sustained supply to those who need it in the frontline. In absence of reliable risk assessment and management based on true incidence calculation leads to either inadequate or overestimation of risk and unjustified use of PPE. The reported global data for occupational risk of COVID -19 for HCW varies greatly but it is reported to be higher than general populations. However, many of these studies has significant limitations, like inadequate risk assessment, community transmission is not accounted or all HCWs not included for analysis.

The investigators propose to conduct a retrospective study to define and quantify the variable occupational and non-occupational risk among various HCWs, to determine the rates of acquisition in the context of level of PPE use and other infection control measures recommended for COVID-19 and also to define the risk of secondary disease transmission to other household members of participants.

ELIGIBILITY:
Inclusion Criteria:

1.2.1 All staffs that are currently working in included hospitals and clinic in 1.2.1.1 Laboratory confirmed positive case- A positive case is where COVID-19 virus is detected through real time polymerase chain reaction (RT PCR) either through oropharyngeal or nasopharyngeal swab which were conducted on HCWs based on national guidelines of UAE and are based on either symptoms, or as part of contact tracing or history of recent international travel.

1.2.1.2 Laboratory confirmed positive case with history of occupational exposure- through contact tracing after an exposure to a known COVID -19 patient in a healthcare setting.

1.2.1.3 Laboratory confirmed positive case with no history of occupational exposure- non-occupational exposures include situations where there was no probable workplace exposure for the healthcare worker, and a community source for the infection through household contact, travel, gathering in public places or visiting to affected area as most likely source of exposure is identified.

Exclusion Criteria:

Staff who refused to participate or withdraw there consent during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Healthcare workers working actively in the included hospitals or clinics and are confirmed positive with COVID-19
Sampling Method: Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Rate of COVID-19 in healthcare workers (HCWs) | 6 months
  Positive HCW divided by total exposed HCWs in that category X 100 Rate will be calculated in 4 different categories.
  1. Front line HCWs (doctors, nurses, respiratory therapist, physiotherapist, dialysis technician, patient assistant etc)
  2. Front line support staffs (Customer care, pharmacist, billing assistance, ambulance driver etc.),
  3. Clinical support staffs- (dietician, food service worker, laundry worker, housekeeping staffs, health record staffs- infection control team etc.)
  4. Non-clinical support staffs- (Administrative support staff.)

SECONDARY OUTCOMES:
clinical severity of infection in HCWs | Within 28 days of illness.
  WHO Ordinal scale
  1. Uninfected No clinical or virological evidence of infection Score 0
  2. Ambulatory : No limitation of activities Score 1, Limitation Score 2.
  3. Hospitalised(Mild disease): No oxygen Score 3, Nasal prongs or Mask Score 4
  4. hospitalised (Severe disease): noninvasive ventilation/high flow nasal canula- score 5, Intubation and mechanical ventilation Score 6, mechanical ventilation and any other oxygen support like vasopressors Score 7
  5. dead score 8

CONTACTS AND LOCATIONS:
Overall Officials: Helen King, RN DMS MBA, Principal Investigator — Senior Vice President: Nursing & Quality Corporate Quality & Nursing
Locations (1):
- NMC Specialty Hospital, Al Nahda, Dubai, United Arab Emirates

REFERENCES:
- [Result] Nguyen LH, Drew DA, Joshi AD, Guo CG, Ma W, Mehta RS, Sikavi DR, Lo CH, Kwon S, Song M, Mucci LA, Stampfer MJ, Willett WC, Eliassen AH, Hart JE, Chavarro JE, Rich-Edwards JW, Davies R, Capdevila J, Lee KA, Lochlainn MN, Varsavsky T, Graham MS, Sudre CH, Cardoso MJ, Wolf J, Ourselin S, Steves CJ, Spector TD, Chan AT. Risk of COVID-19 among frontline healthcare workers and the general community: a prospective cohort study. medRxiv [Preprint]. 2020 May 25:2020.04.29.20084111. doi: 10.1101/2020.04.29.20084111. PMID 32511531
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533